CLINICAL TRIAL: NCT05521997
Title: Phase II Study of Glutaminase Inhibition and Chemoradiation in Advanced Cervical Cancer
Brief Title: Glutaminase Inhibition and Chemoradiation in Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202301163; R01CA181745 (NIH)
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cervical Carcinoma; Cervical Cancer; Cervix Cancer; Cancer of the Cervix
Keywords: advanced cervical cancer; Glutaminase Inhibitor
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Intervention Model Description: Randomization will occur on a 5:1 basis to experimental arm and control arm. The first 5 participants randomized to the experimental arm will be considered the safety lead-in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm: Standard of Care Chemoradiation (Active Comparator): -Participants will receive 7 weeks of standard of care chemoradiation.
  Interventions: Radiation: Radiation treatment; Drug: Cisplatin
- Experimental Arm #1: Telaglenastat + Standard of Care Chemoradiation (Experimental): -Participants will receive 2 weeks of telaglenastat and 7 weeks of standard of care chemoradiation plus telaglenastat.
  Interventions: Drug: Telaglenastat; Radiation: Radiation treatment; Drug: Cisplatin

INTERVENTIONS:
Drug: Telaglenastat — -800 mg twice per day by mouth
  Other Names: CB-893
  Arms: Experimental Arm #1: Telaglenastat + Standard of Care Chemoradiation
Radiation: Radiation treatment — * Standard of care
  * External beam radiation therapy delivered daily 4 days a week and 1 day per week of brachytherapy.
Drug: Cisplatin — * Standard of care
  * Weekly administration of cisplain

SUMMARY:
Advanced cervical cancer patients treated with standard of care (SOC) chemoradiation plus glutaminase inhibition with telaglenastat (CB-839) will have increased progression-free survival (PFS) compared to historical rates for patients receiving SOC chemoradiation alone.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for definitive chemoradiotherapy, including brachytherapy

* Patient age ≥ 18 years.
* Patients with histologically confirmed newly diagnosed advanced cervical cancer (squamous, adenosquamous, adenocarcinoma or poorly differentiated); Federation of Gynecology and Obstetrics (FIGO) 2018 clinical stages III-IVA.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Absolute neutrophil count ≥ 1,500/mcL.
* Platelets ≥ 100,000/mcL.
* Hemoglobin ≥ 8 g/dL (can be transfused prior to study).
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); patients with known Gilbert disease with serum bilirubin ≤ 3 x ULN may be enrolled.
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]/alanine aminotransfersase (ALT) (serum glutamate pyruvate transaminase [SGPT] ≤ 2.5 x ULN.
* Alkaline phosphatase ≤ 2.5 x ULN.
* Serum creatinine ≤ 1.5 mg/dL to receive weekly cisplatin; patients whose serum creatinine is between 1.5 and 1.9 mg/dL are eligible for cisplatin if there is no hydronephrosis and the estimated creatinine clearance (CCr) is ≥ 30 ml/min. For the purpose of estimating the CCr, formulas, including Cockcroft and Gault for females or similar, should be used.
* International normalize ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular weight heparin or warfarin, should be on a stable dose).
* Patient does not have uncontrolled diabetes mellitus (i.e. fasting blood glucose >200 mg/dL).
* Patient does not have a known allergy to cisplatin or compounds of similar biologic composition as CB-839.
* Patient is not actively breastfeeding (or has agreed to discontinue before the initiation of protocol therapy).
* Ability to understand and the willingness to sign a written informed consent document.
* Patients does not have known human immunodeficiency virus syndrome (HIV testing optional).

Exclusion Criteria:

* Patient has another concurrent active invasive malignancy.
* Patient has received prior radiation therapy to the pelvis or previous therapy of any kind for this malignancy, or pelvic radiation for any prior malignancy.
* Patient is receiving another investigational agent for the treatment of cancer.
* Poorly controlled diabetes, with inability to perform 18F-FDG PET scan.
* Patient is pregnant or breastfeeding.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Mean resting QTc > 470 msec obtained by electrocardiogram (ECG).
* Severe, active co-morbidity defined as follows:

  * Current (within 28 days of cycle 1, day 1) signs and/or symptoms of bowel obstruction
  * Patients who require parental hydration and/or nutrition
  * Patients who require drainage gastrostomy tube
  * Evidence of bleeding diathesis or clinically significant coagulopathy
  * Serious, non-healing or dehiscing wound, active ulcer or untreated bone fracture
  * History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month of study enrollment
  * Significant cardiovascular or cerebrovascular disease including: Uncontrolled hypertension (systolic blood pressure [SBP] >= 150; diastolic blood pressure [DBP] >= 90)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2032-03-07 (Estimated); Study Completion 2032-03-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) - experimental arm only | Through completion of follow-up (estimated to be 24 months and 9 weeks)
  * PFS is defined as the duration of time from start of telaglenastat to time of progression or death, whichever occurs first.
  * Progressive disease: New foci of abnormal FDG uptake not present on the pretreatment FDG-PET study

SECONDARY OUTCOMES:
Acute toxicity as measured by number of acute adverse events experienced by participant - experimental arm only | From start of chemoradiation treatment through 90 days
  * Toxicity evaluation will report events according to Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
  * Acute toxicity is defined as any toxicity occurring within 90 days from first receiving study radiotherapy or death, whatever event is observed first.
Late toxicity as measured by number of late adverse events experienced by participant - experimental arm only | From day 91 through 24 months after completion of chemoradiation
  * Toxicity evaluation will report events according to Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
  * Late toxicities include any toxicity that is determined possibly, probably, or definitely related to treatment, within 24 months after completion of treatment.
Overall survival (OS) | Through completion of follow-up (estimated to be 24 months and 9 weeks)
  -OS is defined as the days from the start of Telaglenastat treatment to the date of death, censored at the last follow-up otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Julie K Schwarz, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu